CLINICAL TRIAL: NCT02583581
Title: A Feasibility Study for Examination the Use of Brain Prefrontal Activity Monitoring, for Early Detection of Migraine Attack
Brief Title: Evaluation of Use of Brain Activity Monitoring for Prediction of Migraine Attacks
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brainmarc Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLD4
Record Dates: First submitted 2015-10-01; First posted 2015-10-22 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Participants diagnosed with migraine (Experimental): EEG monitoring (MindWave by NeuroSky and EPOC by Emotiv)
  Interventions: Device: EEG monitoring (MindWave by NeuroSky); Device: EEG monitoring (EPOC by Emotiv)

INTERVENTIONS:
Device: EEG monitoring (MindWave by NeuroSky) — EEG evaluation will be conducted for duration of 10 minutes. 5 minutes without auditory stimulation and 5 minutes with auditory stimulation performed using standard headphone or earphones to reduce external noises.
Device: EEG monitoring (EPOC by Emotiv) — EEG evaluation will be conducted for duration of 10 minutes. 5 minutes without auditory stimulation and 5 minutes with auditory stimulation performed using standard headphone or earphones to reduce external noises.

SUMMARY:
This study evaluates the use of brain activity monitoring for prediction of migraine attacks in an expected time scale of 12-48 hours prior to the migraine attack.

DETAILED DESCRIPTION:
The study will be conducted in one are. Participants diagnosed with migraine, will be evaluated for their EEG characteristics as well as daily migraine related clinical and general status. Participants' monitoring will be conducted for 20 times for a duration of one month.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with migraine by a neurologist.
* Male or Female, aged 18 -50 years.
* Able and willing to comply with all study requirements.
* Having 3-10 migraine attacks per month.

Exclusion Criteria:

* Diagnosed with chronic pain, neurological or psychiatric disorders.
* Current or past use of anti-depressants.
* A user of recreational or illicit drugs or has had a recent history of drug or alcohol abuse or dependence.
* History of seizures
* Head injury with consciousness loss in the last three months.
* Diagnosed as ADHD and/or use of Ritalin.
* Hearing disorder and/or known ear drum impairment.
* Having migraine attacks occurring only during the menstruation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-01 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Measurements of brain electrical signal in Micro volt. | 1 months
  Measurements of brain electrical signal in Micro volt will be quantified by an algorithm and correlated to reported migraine cycle (as reported by migraine patients in questionnaires).

CONTACTS AND LOCATIONS:
Overall Officials: David Yarnitsky, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel